CLINICAL TRIAL: NCT02915289
Title: Chlorhexidine Gluconate vs Povidone-Iodine Vaginal Cleansing Solution Prior to Cesarean Delivery: A Randomized Comparator Controlled Trial
Brief Title: Chlorhexidine Gluconate vs Povidone-Iodine Vaginal Cleansing Solution Prior to Cesarean Delivery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Richmond University Medical Center (Other)
Responsible Party: Principal Investigator, Nisha Lakhi, MD, Director of Research, Richmond University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-08-04 RUMC
Record Dates: First submitted 2016-09-23; First posted 2016-09-27 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Wound Infection; Complication, Postoperative
Keywords: Caesarean section; Chlorhexidine gluconate
MeSH Terms: conditions — Wound Infection; Postoperative Complications | interventions — Povidone-Iodine; chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Povidone Iodine (Active Comparator): 10% povidone iodine solution will be used for vaginal cleansing prior to non-emergent cesarean section. The preparation will be applied according to the manufacture guidelines with a minimum of four completed minutes of drying time before placement of surgical drapes. The group will receive standard obstetrical care, continuous fetal monitoring, and pre-operative prophylactic antibiotics at least one hour prior to skin incision.
  Interventions: Procedure: Povidone Iodine
- Chlorhexidine gluconate (Active Comparator): 4% chlorhexidine gluconate solution will be used for vaginal cleansing prior to non-emergent cesarean section. The preparation will be applied according to manufacture guidelines. The group will receive standard obstetrical care, continuous fetal monitoring, and pre-operative prophylactic antibiotics at least one hour prior to skin incision.
  Interventions: Procedure: Chlorhexidine gluconate

INTERVENTIONS:
Procedure: Povidone Iodine — Vaginal preparation with 10% povidone iodine prior to non-emergent cesarean section.
  Arms: Povidone Iodine
Procedure: Chlorhexidine gluconate — Vaginal preparation with 4% chlorhexidine gluconate prior to non-emergent cesarean section.
  Arms: Chlorhexidine gluconate

SUMMARY:
Endometritis, an infection of the uterus in the postpartum period, has been shown to complicate the postoperative course of a cesarean delivery in 6% to 27% of cases. Vaginal cleansing prior to cesarean delivery has been shown to minimize the presence of micro-organisms and risk of infection. Although povidone-iodine is the most commonly used anti-septic for surgical preparation of the vagina, it is not an ideal agent due to it's diminished efficacy in acidic vaginal pH and in the presence of blood. Chlorhexidine gluconate, on the other hand, has demonstrated superior disinfectant properties in several clinical trials, as compared to povidone iodine. In this randomized, comparator controlled, study the investigators will be comparing chlorhexidine gluconate vs povidone iodine for intrapartum vaginal preparation in women undergoing non-emergent cesarean delivery.

DETAILED DESCRIPTION:
This is a randomized, comparator controlled, study of intrapartum vaginal preparation with either chlorhexidine gluconate or povidone-iodine solution. Women undergoing non-emergent cesarean delivery will be randomized to receive vaginal cleansing with either 4% chlorhexidine solution or 10% providone-iodine solution.

The study will have two arms that will be randomized in a 1:1 ratio. After inclusion criteria have been satisfied, subjects in the comparator control arm will receive vaginal preparation with 10% provodone-iodine solution prior the skin incision. Subjects in the study arm will receive vaginal preparation with chlorohexidine gluconate 4% solution. The selected skin preparation will be applied according to the manufacture guidelines with a minimum of four completed minutes of drying time before placement of surgical drapes. A block randomization method will be used to control for variations in care. Both groups will receive standard obstetrical care, continuous fetal monitoring, and pre-operative prophylactic antibiotics at least one hour prior to skin incision.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Richmond University Medical Center that have a non-emergent cesarean delivery

Exclusion Criteria:

* Emergent cesarean delivery, less than 18 years of age, chorioamnionitis before randomization, intrapartum fever prior to randomization, or known or suspected allergy to chlorhexidine or iodine.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1114 (Actual)
Dates: Start 2016-12; Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Postoperative wound infection | 0-14 days postpartum
  Erythema surrounding the incision site or pus-like incisional drainage in the presence or absence of fever

SECONDARY OUTCOMES:
Postpartum endometritis | 0-14 days post-partum
  Clinical diagnosis with temperature of 100.4 degrees F or higher occurring 24 hours after surgery with uterine fundal tenderness or purulent lochia.
Postoperative fever | 0-14 days post-partum
  Temperature greater than 38 degrees C or 100.4 degrees F
Side effects | 0-14 days post-partum
  Patient reported side effects of vaginal preparation (allergy, irritation)

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Lakhi, MD, Principal Investigator — Richmond University Medical Center
Locations (1):
- Richmond University Medical Center, Staten Island, New York, United States

REFERENCES:
- [Derived] Lakhi NA, Tricorico G, Osipova Y, Moretti ML. Vaginal cleansing with chlorhexidine gluconate or povidone-iodine prior to cesarean delivery: a randomized comparator-controlled trial. Am J Obstet Gynecol MFM. 2019 Mar;1(1):2-9. doi: 10.1016/j.ajogmf.2019.03.004. Epub 2019 Mar 19. PMID 33319753
- [Derived] Haas DM, Morgan S, Contreras K, Kimball S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2020 Apr 26;4(4):CD007892. doi: 10.1002/14651858.CD007892.pub7. PMID 32335895